CLINICAL TRIAL: NCT03531944
Title: The Impact of Community Pharmacist-Involved Collaborative Care in the Management of Primary Care Patients With Type 2 Diabetes Mellitus in Singapore (IMPACT-C)
Brief Title: Impact of Community Pharmacist-Involved Collaborative Care Model for the Management of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Joyce Lee, PharmD, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-18-019
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community pharmacist-involved care (Experimental): Community pharmacist-involved collaborative care in the management of type 2 diabetes mellitus
  Interventions: Other: Community pharmacist-involved collaborative care
- Usual care (Placebo Comparator): Usual care with physician and as needed referral to nurses
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Community pharmacist-involved collaborative care — Community pharmacist-involved collaborative care in the management of individuals with type 2 diabetes mellitus
  Arms: Community pharmacist-involved care
Other: Usual care — Usual care with physician and as needed visit to the nurse
  Arms: Usual care

SUMMARY:
Background: In Singapore, the prevalence of diabetes mellitus was approximately 12.8% in 2014 and the prevalence was projected to rise to 22.7% in 2035. In view of the complexity of diabetes management, collaborative efforts by nurses and other allied health professionals such as dietitians and pharmacists have shown to play a significant role in improving clinical care of individuals with diabetes. Currently in Singapore, the effectiveness of the collaborative care model has only been evaluated prospectively in the primary and tertiary care settings involving clinical pharmacists. The impact of the unique, synergistic roles of community pharmacists with family physician on the clinical, humanistic and economic outcomes have yet to be elucidated.

Aims: This study aims to evaluate the clinical, humanistic, and economic outcomes of a community pharmacist-involved collaborative care model in the management of individuals with type 2 diabetes mellitus.

Hypothesis: Incorporating community pharmacist into the care model with family physician and nurse can improve the clinical, humanistic, and economic outcomes of individuals with type 2 diabetes mellitus.

Methods: This study is a prospective, open label, parallel arm, randomized controlled trial. The study will be conducted over 6 months at a family medicine clinic in Singapore. Individuals aged 21 years and above, diagnosed with type 2 diabetes (HbA1c > 7.0%) and taking 5 or more chronic medications will be eligible. Individuals with Type 1 diabetes or who are unable to communicate independently in English, Mandarin or Malay will be excluded from this study. The participants will be randomly assigned to 2 groups using a random number generator or an equivalent: (1) Usual diabetes care with physician (control), (2) diabetes care with physician and community pharmacist (intervention). The community pharmacist will adopt the core elements of the medication therapy management model in reviewing the medications of participants as well as provide relevant lifestyle counselling and health education via a face-to-face consultation at the clinic and subsequently through telephonic correspondences. The primary outcome will be change in HbA1c over 6 months. Secondary outcomes include blood pressure, lipid markers, distress level, self-care capabilities, quality of life, productivity, and direct medical costs.

Significance: The outcomes of the community pharmacist-involved collaborative care model will support future implementation and integration of this care model into the standard of care in Singapore so as to optimize the management of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* All individuals aged 21 years and above, diagnosed with type 2 diabetes mellitus with a baseline HbA1c of more than 7.0% and taking 5 or more chronic medications

Exclusion Criteria:

* Individuals with type 1 diabetes mellitus
* Mentally incapacitated individuals
* Individuals who are illiterate and unable to communicate in English, Malay, or Chinese (Mandarin)
* Individuals who are not able to complete the questionnaires

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c level | Baseline and 6 months
  Change in HbA1c level over 6 months

SECONDARY OUTCOMES:
Change in blood pressure | Baseline and 6 months
  Change in systolic blood pressure and diastolic blood pressure
Change in lipid markers | Baseline and 6 months
  Change in total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglyceride levels
Change in diabetes-related distress | Baseline and 6 months
  Measured by 20-item Problem Areas in Diabetes (PAID), with each item scoring from 0 to 4. The total score is computed by the sum of score of each item, ranging from 0 to 100 (highest distress level).
Change in general health status | Baseline and 6 months
  Measured by EuroQoL 5-Dimension 5-Level (EQ-5D-5L), each item scored individually on a scale of 1 to 5 (1 being least problem and 5 being most problem). EQ-5D-5L comes with a visual analogue scale assessing general health-related quality of life on that day, ranging from 0 (worst health imaginable) to 100 (best health imaginable).
Change in diabetes-specific quality of life | Baseline and 6 months
  Measured by the 21-item Audit of Diabetes-Dependent Quality of Life (ADDQoL), with 2 global general quality of life questions and 19 domains with weighted score between impact and importance. The average weighted impact is the average of the impact of all domains (ranging from -9, being worst quality of life to +3, being best quality of life).
Change in general work productivity | Baseline and 6 months
  Measured by 6-item Work Productivity Activity Impairment-Global Health (WPAI-GH), four primary outcomes based on the questions including:
  Per cent of work time missed due to health conditions (absenteeism): Q2/(Q2+Q4).
  Per cent impairment while working due to health conditions (presenteeism): Q5/10.
  Per cent overall work impairment due to health: Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))×(Q5/10)].
  Per cent impairment in activities due to health: Q6/10.
Change in self efficacy and self-care capabilities | Baseline and 6 months
  Measured by Summary of Diabetes Self-Care Activities scale (SDSCA),comprised of items assessing five domains of diabetes self-management which are "general diet (2 items), specific diet (2 items), exercise (2 items), blood glucose testing (2 items) and foot care (2 items) and the medication self-management component and smoking self-management component. Each item will be reported as a mean across the sample and analysed individually.
Incidence of hypoglycemia | Baseline and 6 months
  Incidence of hypoglycemia over 6 months
Cost effectiveness analysis | 6 months
  Cost effectiveness of the community pharmacist-involved collaborative care model

CONTACTS AND LOCATIONS:
Locations (1):
- Keat Hong Family Medicine Clinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lum ZK, Tan JY, Wong CSM, Kok ZY, Kwek SC, Tsou KYK, Gallagher PJ, Lee JY. Reducing economic burden through split-shared care model for people living with uncontrolled type 2 diabetes and polypharmacy: a multi-center randomized controlled trial. BMC Health Serv Res. 2024 Jun 22;24(1):760. doi: 10.1186/s12913-024-11199-2. PMID 38907254